CLINICAL TRIAL: NCT04078256
Title: EFFECTIVENESS OF A PROPRIOCEPTIVE EXERCISE PROGRAM IN THE PREVENTION OF INJURIES IN RECREATIONAL RUNNERS
Brief Title: The Importance of Exercise to Prevent Injuries in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/HU/2018/29
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Injury;Sports
Keywords: proprioception; running; prevention; injuries
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group will carry out the proprioceptive exercise program during 8 weeks at the begining of the season
  Interventions: Other: Proprioceptive exercise program
- Control group (Placebo Comparator): Control group will continue with their usual training routine
  Interventions: Other: Usual training routine

INTERVENTIONS:
Other: Proprioceptive exercise program — Group A will carry out two sessions of proprioceptive training per week, in a total of 8 weeks, during the pre-season period (September-October). Each session will last approximately 30 minutes and will include 6 exercises. The execution of the exercises will be supervised by a physiotherapist and a national trainer of athletics.
  Arms: Experimental group
Other: Usual training routine — The subjects of the control group (group B) will be informed so that they do not include any change in their usual training routine.
  Arms: Control group

SUMMARY:
Introduction: running is one of the most accessible and practiced sports in the world since the 21st century. Unfortunately, the incidence of injuries in the population that practices it is high regardless of experience, although the risk of injury increases in amateur runners. One of the main keys to reduce the incidence of running related injuries may be to improve the ability to reduce the load or impact. For this, there are different strategies such as a gradual increase in the load to run, and exercise within which is muscle strengthening and balance training or proprioception.

Objective: to verify the effectiveness of a program of proprioceptive exercises based on the static and dynamic balance for the reduction of lower limb injuries in amateur runners during the competition season.

DETAILED DESCRIPTION:
Methodology: 66 amateur runners, after simple size calculation, will be randomized into two groups. Experimental group will carry out the proprioceptive exercise program during 8 weeks at the begining of the season and control group will continue with their usual training routine. The main variable running related injury will be collected weekly during the follow-up.

Results: When all the data needed for the study has been collected, researchers gathers results and exports them for statistical interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Weekly training of at least 15 kilometers.
* At least practice running 6 months for 1-3 times a week.

Exclusion Criteria:

* To have some type of lower limb or lower back injury at present or in the last 6 months.
* Having undergone surgery for any back or lower limb injury.
* Pregnant.
* Neural dysfunction / disability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Knee Joint Position Sense (JPS) | Change from Baseline Joint Position Sense Pressure at 8 weeks
  JPSThe JPS is defined as the awareness of the actual position of the limb to quantify proprioception.The method for measuring JPS is to place the joint at a specific target angle and then, after the limb has been moved back to the starting angle, the subject is asked to actively or passively reproduce the target angle. The outcome of the measurement is the absolute error (AE), which is the difference between the true target angle and the reproduced angle

SECONDARY OUTCOMES:
The Y Balance Test (YBT) | Change from Baseline dynamic balance at 8 weeks
  The YBT, derived from the Star Excursion Balance Test (SEBT), has been reported to be a valid and reliable measure of dynamic balance; furthermore, the results of the YBT have been reported to be related to lower-extremity impairments and to be predictors of injuries.The YBT instrument has a central raised platform with three pieces of PVC (polyvinyl chloride) pipe in the three directions with a sliding plastic reach indicator that the participant pushes to determine reach distance.The YBT testing protocol assessed absolute reach and normalized distance for each direction, asymmetry between limbs, and composite score. Normalized reach distance is calculated by dividing reach distance by the limb length. Asymmetry is the absolute difference between right and left leg and is determined for each reach direction. The composite score is calculated by summing the reach distance in the three directions, dividing by three times limb length, and multiplying by 100.
The countermovement jump (CMJ) | Change from Baseline jump height at 8 weeks
  The CMJ is primarily used to measure an athlete's explosive lower-body power, and has become one of the most frequently used tests by coaches and researchers to indirectly measure power in the lower limbs. CMJ performance is reported as either jump height(centimeters).

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, Dr., Study Chair — Alcala University
Locations (1):
- Grupo Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain